CLINICAL TRIAL: NCT03317951
Title: A Randomized Controlled Trial for Investigating a Novel Integrated Care Concept (NICC) for Patients Suffering From Chronic Cardiovascular Disease: CardioCare MV
Brief Title: Investigation of a Novel Integrated Care Concept (NICC) for Patients Suffering From Chronic Cardiovascular Disease
Acronym: CardioCare MV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Rostock (Other)
Collaborators: AOK Nordwest (Industry); Techniker Krankenkasse (Other); Philips GmbH Market DACH (Unknown); AMEDON GmbH (Unknown); Lohfert & Lohfert AG (Unknown); Society for Network & Innovation Management of Industry (Germany) (Other); Gemeinsamer Bundesausschuss (Unknown); Universitätsmedizin Rostock Versorgungsstrukturen GmbH (Unknown)
Responsible Party: Principal Investigator, Christian Schmidt, Ärztlicher Vorstand, University of Rostock
Organization: University of Rostock (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2017-0117
Record Dates: First submitted 2017-10-05; First posted 2017-10-23 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure; Atrial Fibrillation; Treatment Resistant Hypertension
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, open-label, randomized, bicenter study parallel-group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel integrated care concept (NICC) (Experimental): The care center is at the heart of the NICC structure. It will be available 24/7. It is the core platform to share information for all NICC patients in the care process and serves as integration point between the professional groups. The care center is utilizing the NICC platform for care coordination and patient monitoring. The NICC platform enables patient management from the distance and allows treating physicians to observe and follow the health status of patients daily. Using the NICC tablet, patients provide information from home about their health status. They will receive feedback about their therapy, measurements and reminders and motivation to follow care plans. The communication allows for a regular evaluation of the patient's situation, a review of the therapy and coordination of necessary adjustments with care providers. The general intervention rules are based on the current European Society of Cardiology (ESC) guidelines for treating AF, HF and TRH patients.
  Interventions: Other: Novel integrated care concept (NICC)
- Standard care (Active Comparator): Patients will be treated according to current practice as described in the guidelines of the European Society of Cardiology (ESC). For AF, this has been provided by Kirchhof et al. (2016 Eur Heart J). HF treatment will follow the 2016 ESC guideline for HF (Ponikowski et al., 2016 Eur Heart J), and TRH will be treated according to the ESC treatment guideline for arterial hypertension (Mancia et al., 2013 Eur Heart J).
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Novel integrated care concept (NICC) — Integrated care concept including, e.g., call center, guideline therapy, tablet and medical devices
  Arms: Novel integrated care concept (NICC)
Other: Standard care — Guideline therapy according to the guidelines of the European Society of Cardiology (ESC).
  Arms: Standard care

SUMMARY:
Cardiovascular diseases are the number 1 cause of death globally and represent a major economic burden on health care systems. The investigators have developed a novel integrated care concept (NICC) which combines telemedicine with intensive support by a call center, an integrated care network including in- and outpatient care providers and guideline therapy for patients with heart failure (HF), atrial fibrillation (AF) or therapy resistant hypertension (TRH). The aim of the study is to show that NICC is preferable over guideline therapy alone. We aim at including approximately 890 patients. Patients could be enrolled either directly at the Care-Center (location: University Hospital of Rostock) or at one of the advanced treatments rooms of the Care-Center (outpatient cardiological specialist practices).

The ethics commission's statement of the University of Rostock is available for amendment 2 since 20.08.2019 at the number A2017-0117.

DETAILED DESCRIPTION:
Background: Cardiovascular diseases are the number 1 cause of death globally and represent a major economic burden on health care systems. Positive effects of disease management programs have been shown for patients with heart failure (HF). Remote monitoring and telemonitoring with active intervention are beneficial in atrial fibrillation (AF) and therapy resistant hypertension (TRH), respectively. For these patients, the investigators have developed a novel integrated care concept (NICC) which combines telemedicine with intensive support by a call center, an integrated care network including in- and outpatient care providers and guideline therapy for patients.

Methods: The aim of the study is to demonstrate the superiority of NICC over guideline therapy alone. The trial is designed as open-label bi-center parallel-group design with two groups. Patients will be included if they are either inpatients or if they are referred to the outpatient clinic of the hospitals by their treating physician. Randomization will be done individually with stratification by cardiovascular disease (AF, HF, TRH), center and admission type. Primary endpoints are based on the 1-year observation period after randomization. The first primary endpoint is the composite endpoint consisting of mortality, stroke and myocardial infarction. The number of hospitalizations form the second primary endpoint. The third primary endpoint is identical to the first primary endpoint plus cardiac decompensation. Adjustments for multiple testing are done using a fall back strategy. Secondary endpoints include patient adherence, health care costs, quality of life and safety. The power for the second primary endpoint is 80% at the two-sided 2.5% test-level with a sample size of 890 patients.

Discussion: This study will inform care providers whether quality of care can be improved by an integrated care concept providing telemedicine through a 24/7 care center approach. We expect that cost of the NICC will be lower than standard care because of reduced hospitalizations. If the study has a positive result, NICC is planned to be immediately rolled out in the state of Mecklenburg-West Pomerania. The trial will also guide additional research to disentangle the effects of this complex intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Heart failure (I50, NYHA II-IV) or atrial fibrillation (I48, EHRA II-IV) or resistant hypertension (I10-15, ≥ 3 antihypertensive medicines from different drug classes, SBP > 140 /90mmHg or ≥ 4 antihypertensives irrespective of the blood pressure, with at least one drug being a diuretic).
2. Member of health insurance company AOK Nordost or Techniker Krankenkasse (TK).
3. Inscription to integrated care contract with the health insurance company.
4. Residence in Mecklenburg-Vorpommern.
5. Age ≥ 18 years.
6. Written informed consent.

Exclusion Criteria:

1. Pregnancy, suspected pregnancy or breast-feeding period.
2. Participation in another clinical trial up to 30 days before inclusion in this trial.
3. Cognitive deficits: patients need to be able to read and understand German language as presented on a tablet.
4. Chronic kidney disease requiring dialysis or creatinine clearance < 15 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint death and cardiovascular events | 1-year after randomization
  Composite endpoint consisting of mortality (occurrence: yes/no), stroke (yes/no) and myocardial infarction (yes/no) within the 1-year observation period. Endpointed rated as yes if at least one yes
Hospitalization | 1-year after randomization
  Number of hospitalizations within the 1-year observation period
Composite endpoint death and broader cardiovascular events | 1-year after randomization
  Composite endpoint consisting of mortality (occurrence: yes/no), stroke (yes/no), myocardial infarction (yes/no) and cardiovascular decompensation (yes/no) within the 1-year observation period. Endpointed rated as yes if at least one yes.

SECONDARY OUTCOMES:
Adherence to novel integrated care concept | 1-year after randomization
  Adherence to novel integrated care concept as measured, e.g., as percent of completed blood pressure measurements in patients with blood pressure device.
Quality of life | Baseline, 6 months, 1 year
  Change in EuroQol (EQ-5D-5L). EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, will be converted into a single index value. The EQ-5D-5L index value will be calculated using the Crosswalk Index Value Calculator based on data from the German population. EQ-5D-5L analyses will be done separately for each level and each category.
Cost | 1-year after randomization
  Treatment cost within the 1-year observation period
Safety as measured by cardiovascular events | 1-year after randomization
  Mortality, stroke, TIA, myocardial infarction, hospitalization, cardiovascular decompensation. All measured as yes/no within the 1-year observation period.
Beliefs about medicine questionnaire | Baseline, 6 months, 1 year
  The BMQ consists of two sections, general and specific. The specific section assesses patients' beliefs about medications prescribed for a particular illness. Each statement has a 5-point Likert scale answers with 1 = strongly disagree, 2 = disagree, 3 = uncertain, 4 = agree and 5 = strongly agree. Points of each scale are summed to give a scale score. Higher scores indicate stronger beliefs in the concepts of the scale.
Time to event | 1-year after randomization
  Primary composite endpoints as time to event
Medication adherence report scale | Baseline, 6 months, 1 year
  Self-reported adherence will be assessed using the MARS-5. Respondents score on 5-point Likert scales. The first statement of the MARS asks patients about unintentional non-adherence, whereas the other 4 statements question intentional non-adherence. The total score ranges from 5 to 25, with higher scores indicating higher self-reported adherence.
Illness-specific Social Support Scale Short version-8 | Baseline, 6 months, 1 year
  The 8-item version of the ISSS measures positive support and detrimental interaction with four items each. Items are scored on a 5-point Likert scale ranging from 0 ('never') to 4 ('always'), and total scores may therefore range from 0 to 16.
Patient activation measure | Baseline, 6 months, 1 year
  The PAM13-D is an interval level, unidimensional Guttman-like scale with items sequenced by difficulty of activation. Patient activation is measured on a 0-100 scale, and activation scores can be converted to a four-level category score as described by Insignia Health.
Heart specific quality of life | Baseline, 6 months, 1 year
  The HeartQoLis a health-related quality of life questionnaire with 14 items.The 14-items in the HeartQoL scale cluster as a 10-item physical and a 4-item emotional subscale. Items score from 0 to 3 on a Likert scale, and means are calculated for each of the two domains and the total score. Higher scores indicate better quality of life.
Patient Health Questionnaire depression module | Baseline, 6 months, 1 year
  The PHQ-9 is the WHO depression module, which scores each of the 9 diagnostic criteria for major depression in Diagnostic and Statistical Manual Fourth Edition using a 4-point Likert scale which are 0 "not at all," 1 "several days," 2 "more than half the days" and 3 "nearly every day". Total scores may therefore range from 0 to 27.
Generalized Anxiety Disorder scale | Baseline, 6 months, 1 year
  The GAD-7 assesses the most prominent diagnostic features (diagnostic criteria A, B, and C from the Diagnostic and Statistical Manual of Mental Disorders, fourth edition [DSM-IV]) for GAD. Items are scored on a 4-point Likert scale, and they are 0 "not at all," 1 "several days," 2 "more than half the days" and 3 "nearly every day". The total score therefore ranges from 0 to 21. Low values represent no or mild anxiety.
World Health Organization Well-Being Index | Baseline, 6 months, 1 year
  The 5-item WHO Well-Being Index (WHO-5) assesses subjective psychological well-being.The respondent is asked to rate how well each of 5 statements applies to him or her when considering the last 14 days. Items are scored on a 6-point Likert scale from 5 "all of the time" to 0 "none of the time". The raw sum score ranges from 0, absence of well-being, to 25, maximal well-being. The scores are multiplied by 4 for a transformation to a percentage scale with values from 0 "absent" to 100 "maximal".

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schmidt, Prof Dr, Principal Investigator — Universitätsmedizin Rostock
Locations (1):
- Universitätsmedizin Rostock, Rostock, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oner A, Dittrich H, Arslan F, Hintz S, Ortak J, Brandewiede B, Mann M, Krockenberger K, Thiery A, Ziegler A, Schmidt C; CardioCare MV Study Group. Comparison of telemonitoring combined with intensive patient support with standard care in patients with chronic cardiovascular disease - a randomized clinical trial. Eur J Med Res. 2023 Jan 11;28(1):22. doi: 10.1186/s40001-023-00991-1. PMID 36631889
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Ziegler A, Mann M, Brandewiede B, Dittrich H, Hintz S, Krockenberger K, Oner A, de Sousa MO, Schmidt C. Statistical analysis plan for the randomized controlled trial CardioCare MV investigating a novel integrated care concept (NICC) for patients suffering from chronic cardiovascular disease. Trials. 2020 Feb 3;21(1):131. doi: 10.1186/s13063-020-4052-6. PMID 32014033
- [Derived] Schmidt C, Oner A, Mann M, Krockenberger K, Abbondanzieri M, Brandewiede B, Bruge A, Hostenkamp G, Kaiser A, Neumeyer H, Ziegler A. A novel integrated care concept (NICC) versus standard care in the treatment of chronic cardiovascular diseases: protocol for the randomized controlled trial CardioCare MV. Trials. 2018 Feb 20;19(1):120. doi: 10.1186/s13063-018-2502-1. PMID 29458404